CLINICAL TRIAL: NCT00234520
Title: A Multicentre Prospective Controlled Observer Blinded Cohort Study in Patients With Acromegaly to Evaluate the Risk of Cardiac Valvular Regurgitation in Patients Treated With Lanreotide Relative to Patients Treated With Octreotide
Brief Title: A Study to Evaluate the Risk of Developing a Heart Condition Called Valvular Regurgitation in Patients With Acromegaly Treated With Either Lanreotide or Octreotide
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: 2-47-52030-721
Record Dates: First submitted 2005-10-05; First posted 2005-10-07 (Estimated); Last update posted 2019-08-02 (Actual); Status verified 2019-08

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The aim of the study is to compare the risk of acromegaly patients developing valvular regurgitation when receiving lanreotide or octreotide

ELIGIBILITY:
Inclusion Criteria:

* Patient has a diagnosis of Acromegaly
* Patient is being treated with lanreotide or octreotide in any dose form at the selection visit or is a de novo patient who is due to commence treatment within 2 weeks of baseline
* Patient started treatment with either lanreotide or octreotide when both products were available on the market in their country
* Patient must not change treatment form lanreotide to octreotide or vice versa for the duration of the study

Exclusion Criteria:

* Patients with known significant valve abnormalities prior to treatment with either lanreotide or octreotide
* Patients who have received treatment with a somatostatin analogue other than lanreotide or octreotide for more than 3 months
* Patients who have received treatment with a GH antagonist for more than 3 months
* Patients who have had heart valve replacement therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2003-05; Primary Completion 2005-02-18 (Actual); Study Completion 2005-02-18 (Actual)

PRIMARY OUTCOMES:
Assessment of the risk of new or worsening valvular regurgitation in any valve by echocardiography at baseline & 12 months

SECONDARY OUTCOMES:
Assessment of the risk of new or worsening valvular regurgitation in any valve by echocardiography at baseline & 6 months
Risk in each of the 4 valves at 6 & 12 months
Risk of significant regurgitation in each valve at 6 & 12 months
Prevalence of valvular regurgitation at baseline
Assessment of GH and IGF-1 levels at baseline, 6 months & 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (33):
- Belgium (3):
  - Cliniques Universitaires Saint Luc, Brussels
  - UZ Gasthuisberg, Leuven
  - CHU de Liege, Liège
- Czechia (2):
  - University Hospital, Charles University, Kralove
  - 1st School of Medicine, Charles University, Prague
- National University Hospital, Copenhagen, Denmark
- France (7):
  - Hôpital de Bois, Bois-Guillaume
  - Hôpital de la Timone, Marseille
  - CHU de Brabois, Nancy
  - Centre Hospitalier Régional d'Orléans, Orléans
  - Hôpital du Haut-Lévêque, Pessac
  - Hôpital Maison Blanche, Reims
  - CHU de Rangueil, Toulouse
- Hungary (2):
  - Semmelweis University Medical School, Budapest
  - National Medical Center, Budapest
- Italy (6):
  - Ospedali Riuniti di Bergamo, Bergamo
  - Università degli Studi di Ferrara, Ferrara
  - Dipartimento di Scienze, Endocrinologiche e Metaboliche, Genova
  - Università degli Studi di Milano, Milan
  - University "Federico II" of Naples, Naples
  - Clinica Medica II, Roma
- Bielanski Hospital, Warsaw, Poland
- Spain (3):
  - Hospital General de Alicante, Alicante
  - Clínica Puerta de Hierro, Madrid
  - Fundación Jiménez Díaz, Madrid
- Sweden (3):
  - Research Centre for Endocrinology and Metabolism, Gothenburg
  - Endokrinologiska kliniken, Malmo
  - Karolinska Sjukhuset, Stockholm
- United Kingdom (5):
  - Queen Elizabeth Medical Centre, Edgbaston, Birmingham
  - Royal Free Hospital, Hampstead
  - Michael White Diabetes Centre, Hull
  - Christie Hospital, Manchester
  - Northern General Hospital, Sheffield

REFERENCES:
- [Result] Colao A, Marek J, Goth MI, Caron P, Kuhn JM, Minuto FM, Weissman NJ. No greater incidence or worsening of cardiac valve regurgitation with somatostatin analog treatment of acromegaly. J Clin Endocrinol Metab. 2008 Jun;93(6):2243-8. doi: 10.1210/jc.2007-2199. Epub 2008 Apr 1. PMID 18381583